CLINICAL TRIAL: NCT00309491
Title: A Randomized Phase III Study Comparing Tamoxifen vs. Tamoxifen + Aminoglutethimide in Postmenopausal, Hormone Receptor-positive Patients
Brief Title: Randomized Study Comparing Tamoxifen vs. Tamoxifen + Aminoglutethimide in Postmenopausal Receptor-positive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABCSG-6
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Early-stage Breast Cancer
Keywords: Tamoxifen; Aminoglutethimide; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Aminoglutethimide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (Experimental): Tamoxifen alone
  Interventions: Drug: Tamoxifen alone
- Group II (Experimental): Tamoxifen + Aminoglutethimide
  Interventions: Drug: Tamoxifen alone; Drug: Tamoxifen + Aminoglutethimide

INTERVENTIONS:
Drug: Tamoxifen alone — 2 x 20 mg tamoxifen daily, start of therapy within 4 weeks after surgery; therapy duration 5 years
  Other Names: Nolvadex
Drug: Tamoxifen + Aminoglutethimide — 2 x 20 mg tamoxifen daily (5 years) plus Aminoglutethimide daily (first 2 years)
  * 1st therapy week:125mg/-/125mg Aminoglutethimide daily
  * 2nd therapy week: 125mg/-/250mg Aminoglutethimid daily
  * as of 3rd therapy week: 250mg/-/250mg Aminoglutethimid daily
  Other Names: Nolvadex + Orimeten
  Arms: Group II

SUMMARY:
Primarily, this clinical investigation compared the efficacy of tamoxifen + aminoglutethimide vs. tamoxifen alone in terms of prognosis (overall survival) in postmenopausal patients with potentially curative, operated hormone receptor-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal patients with histologically verified, locoradically treated, invasive or minimally invasive breast cancer
* Hormone receptor-positive status
* More than 6 histologically examined lymph nodes
* Laboratory parameters

  1. hematopoiesis: > 3500/µl leucocytes, > 100,000/µl thrombocytes
  2. renal function: creatinin < 1.5mg%
  3. hepatic function: GOT < 2.5 x UNL
  4. bilirubin: < 1.5mg %
  5. metabolic parameters: Na, Ca, K in normal range, normal level of blood sugar
* Concluded healing process following surgery
* Less than 4 weeks interval since surgery
* Informed consent

Exclusion Criteria:

* Premenopausal patients, non-determinable menopausal status
* Previous radiotherapy, chemotherapy or endocrine treatment
* Generalized disease (as verified by lung X-ray, skeletal X-ray, liver ultrasound)
* Contraindications against tamoxifen or anastrozole
* T4 tumors; carcinoma in situ
* Lacking compliance or understanding of disease
* Karnofsky Index < 3
* Serious concomitant disease
* Septic complications, systemic infections or infectious local processes
* Bilateral ovariectomy or ovarian irradiation
* Second carcinoma or status post second carcinoma (except for treated squamous cell carcinoma of the skin or cervical carcinoma in situ)

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2021 (Actual)
Dates: Start 1990-12 (Actual); Primary Completion 1996-01 (Actual); Study Completion 2000-03 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Recurrence-free survival
Side-effect profiles

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Jakesz, MD, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pfeiler G, Stoger H, Dubsky P, Mlineritsch B, Singer C, Balic M, Fitzal F, Moik M, Kwasny W, Selim U, Renner K, Ploner F, Steger GG, Seifert M, Hofbauer F, Sandbichler P, Samonigg H, Jakesz R, Greil R, Fesl C, Gnant M; ABCSG. Efficacy of tamoxifen +/- aminoglutethimide in normal weight and overweight postmenopausal patients with hormone receptor-positive breast cancer: an analysis of 1509 patients of the ABCSG-06 trial. Br J Cancer. 2013 Apr 16;108(7):1408-14. doi: 10.1038/bjc.2013.114. Epub 2013 Mar 19. PMID 23511562
- [Background] Schmid M, Jakesz R, Samonigg H, Kubista E, Gnant M, Menzel C, Seifert M, Haider K, Taucher S, Mlineritsch B, Steindorfer P, Kwasny W, Stierer M, Tausch C, Fridrik M, Wette V, Steger G, Hausmaninger H. Randomized trial of tamoxifen versus tamoxifen plus aminoglutethimide as adjuvant treatment in postmenopausal breast cancer patients with hormone receptor-positive disease: Austrian breast and colorectal cancer study group trial 6. J Clin Oncol. 2003 Mar 15;21(6):984-90. doi: 10.1200/JCO.2003.01.138. PMID 12637461
- [Background] Rudas M, Lehnert M, Huynh A, Jakesz R, Singer C, Lax S, Schippinger W, Dietze O, Greil R, Stiglbauer W, Kwasny W, Grill R, Stierer M, Gnant MF, Filipits M; Austrian Breast and Colorectal Cancer Study Group. Cyclin D1 expression in breast cancer patients receiving adjuvant tamoxifen-based therapy. Clin Cancer Res. 2008 Mar 15;14(6):1767-74. doi: 10.1158/1078-0432.CCR-07-4122. PMID 18347178
- [Derived] Wimmer K, Hlauschek D, Balic M, Pfeiler G, Greil R, Singer CF, Halper S, Steger G, Suppan C, Gampenrieder SP, Helfgott R, Egle D, Filipits M, Jakesz R, Solkner L, Fesl C, Gnant M, Fitzal F. Is the CTS5 a helpful decision-making tool in the extended adjuvant therapy setting? Breast Cancer Res Treat. 2024 Jun;205(2):227-239. doi: 10.1007/s10549-023-07186-6. Epub 2024 Jan 25. PMID 38273214
- See also: Click here for more information about this study: publications — http://www.abcsg.at